## Preschooler Emotion Regulation in the Context of Maternal Borderline Personality Disorder Statistical Analysis Plan NCT03060902

April 11, 2023

We conducted preliminary analyses to examine descriptive statistics by maternal group status (randomly assigned to DBT Skills vs Family Services as Usual) and bivariate correlations between all study variables using IBM SPSS Statistics (Version 26.0). In addition, we examined the extent to which our RCT produced change in maternal ER difficulties using Repeated Measures ANOVA. Maternal emotion regulation was measured using the Difficulties in Emotion Regulation Scale, across all 4 time points.

All primary analyses were conducted in MPlus version 8 (Muthén & Muthén, 2017) using full information maximum likelihood with robust standard errors (MLR) to handle missing data. Model fit was evaluated using standard criteria for chi-square, comparative fit index (CFI; Bentler, 1990), and the root mean square error of approximation (RMSEA, Browne & Cudeck, 1993).